CLINICAL TRIAL: NCT04135534
Title: Find the Adequate Dose of Nalbuphine for Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, KMUHIRB-F(I)-20190070, Principal Investigator, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20190070
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Post Operative Pain; Opioid Side Effects
Keywords: nalbuphine dose
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (Active Comparator): mutonpain 0.05 mg/kg
  Interventions: Drug: group A
- Group B (Active Comparator): mutonpain 0.1 mg/kg
  Interventions: Drug: group B
- Group C (Active Comparator): mutonpain 0.2 mg/kg
  Interventions: Drug: group C

INTERVENTIONS:
Drug: group A — mutonpain 0.05 mg/kg
  Arms: group A
Drug: group B — mutonpain 0.1 mg/kg
  Arms: Group B
Drug: group C — mutonpain 0.2 mg/kg
  Arms: Group C

SUMMARY:
This study evaluate the adequate dose of mutonpain for laparoscopic cholecystectomy in the management of post operative pain. The investigators will randomize patients into three groups to compare the analgesia effects and side effects.

DETAILED DESCRIPTION:
Nalbuphine is a FDA approved noncontrolled drug of opioid. And it had been applied for post operative pain for different surgeries, claiming that less nausea and vomiting with the same analgesic effect when comparing with morphine.

However, several studies concerning post pain management usually used nalbuphine 0.15-0.3 mg/kg for laparoscopic cholecystectomy. If the analgesic effect of nalbuphine is similar with morphine, less nalbuphine injection could reduce the side effects of opioid.

The investigators will randomize patients into three groups of different initial nalbuphine dose for post laparoscopic cholecystectomy surgical pain, and set patient control analgesia machine with nalbuphine for further pain management. If the pain or side effects of opioid were intolerable, the investigators will change pain medications into NSAIDs or other adequate medications to comfort the patient.

The primary outcome were numerical rating pain score and consumption of nalbuphine. The secondary outcomes were nausea, vomiting, pruritus and satisfactory score, and if any other medications use.

ELIGIBILITY:
Inclusion Criteria:

* patient accept laparoscopic cholecystectomy
* age:20-80 years old

Exclusion Criteria:

* nalbuphine allergy
* chronic pain
* active liver disease that would affect metabolization of nalbuphine
* patient who had regular pain medications
* patient who could not cooperate to the evaluation of the survey
* dementia or other psychiatric disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Pain Scale | numerical rating pain scale change at post-operative 1 hour, 2 hours, 4 hours, 24 hours, 36 hours
  The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). The investors will measure the pain score at rest state and upon movement state at post-operative 1 hour, 2 hours, 4 hours, 24 hours, 36 hours.
consumption of nalbuphine | Record the opioid dose changes 2 days.
  The investors will use patient control analgesia machine to calculate the time dependent dose of nalbuphine.

SECONDARY OUTCOMES:
nausea | the nausea sensation changes at post operation 1 hour, 2 hours, 4 hours, 24 hours, 36 hours
  we will go to bed side and have an self-report episode of nausea at 1 hour, 2 hours, 4 hours, 24 hours, 36 hours post operation
vomiting | the vomiting episodes at post operation 1 hour, 2 hours, 4 hours, 24 hours, 36 hours
  we will go to bed side and have an self-report episode of vomiting at 1 hour, 2 hours, 4 hours, 24 hours, 36 hours post operation
satisfactory score by net promoter score | 2 days
  The net promoter score is a subjective measure in which individuals rate their satisfactory on an ten-point numerical scale. The scale is composed of 1 to 10. We will measure the net promoter score at the end of the study
use of rescue pain medications | record if any rescue pain medications at post operation 1 hour, 2 hours, 4 hours, 24 hours, 36 hours
  if the patient use other pain medication on request of poor pain control or poor tolerant of the side effects of nalbuphine

OTHER OUTCOMES:
use of antiemetics | 2 days
  if the patient use of antiemetics during the hospitalization
use of antipruritics | 2 days
  if the patient use of antipruritics during the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Guan-Yu Chen, MD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan